CLINICAL TRIAL: NCT00476567
Title: Training During Pregnancy - Effects of Regular Exercise During Pregnancy in Prevention of Pregnancy-related Diseases and Complications During Labour. A Randomised Clinical Trial
Brief Title: Effects of Regular Exercise During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REK4.2007.81
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Pregnancy Complications
Keywords: exercise; pregnancy; prevention; pregnancy-related diseases; labor; complications; physiotherapy
MeSH Terms: conditions — Pregnancy Complications; Motor Activity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise (Experimental): Regular exercise 45-60 minutes minimum three times per week
  Interventions: Behavioral: specific training program
- control (Active Comparator): standard antenatal care
  Interventions: Other: standard

INTERVENTIONS:
Other: standard — standard antenatal care
  Arms: control
Behavioral: specific training program — a specific training program 12 weeks between pregnancy week 20 and 36. regular exercise 45-60 minutes minimum three times per week.
  Other Names: physiotherapy; regular training; specific exercises
  Arms: exercise

SUMMARY:
There is a great lack of results from randomized clinical trials with high methodological quality, assessing the effects of exercise during pregnancy. The main aims of this trial is to study the effects of exercise during pregnancy in the prevention and treatment of disease and complications which may arise during pregnancy:

* Does regular exercise during pregnancy aid in preventing gestational diabetes?
* Does regular exercise during pregnancy prevent low back and/or pelvic girdle pain?
* Does regular exercise during pregnancy prevent urine and/or fecal incontinence?
* Does regular exercise during pregnancy have an effect on labour and delivery?
* Does regular exercise during pregnancy prevent maternal excessive weight gain and fetal macrosomatia?

DETAILED DESCRIPTION:
Pregnancy is regarded as a period of high risk when it comes to development of e.g. excessive weight gain, gestational diabetes and musculoskeletal problems such as low back pain and pelvic girdle pain, and urinary and fecal incontinence. While pregnancy and labor imply these and other risks, exercise is regarded as advantageous during pregnancy. Today's knowledge about the importance of exercise during pregnancy is mainly based on observational data from epidemiological studies, and the scientific strength of the clinical recommendations given is open to question. There is a great lack of results from randomized clinical trials with high methodological quality, assessing the effects of exercise during pregnancy. As a result of this, many important questions are still not answered. One of these is the effect exercise during pregnancy has in the prevention and treatment of disease and complications which may arise during pregnancy. Another question is the consequences that exercise during pregnancy has for labor and delivery. This study is designed as a randomized clinical trial using validated measurement tools to find answers to the mentioned questions.

In both national and international literature the importance of physical activity is highlighted. WHO has recently presented a global strategy for nutrition, physical activity and health. In Norway physical activity and exercise have been strongly addressed, and is an issue of high priority also in pregnant and postpartum women (St.meld.nr.16). Nevertheless, few trials evaluating the effects of regular exercise have been published. There is a need for evidence based knowledge to be implemented in education of health professionals, and in the development of health promotion strategies aiming at the general population.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant 18 weeks
* attend the routine ultrasound control at the three hospitals
* healthy
* age 18 years or more
* singleton live foetus at the routine ultrasound scan
* normal pregnancy.

Exclusion Criteria:

* pregnancy complications
* high risk for preterm labour
* pain during pelvic floor muscle contractions
* ongoing urinary tract infection
* diseases that could interfere with participation (following recommendations from SEF 2000, ACOG 2003)
* living too far from the hospitals to be able to attend weekly exercise groups

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 855 (Actual)
Dates: Start 2007-05; Primary Completion 2011-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Gestational diabetes | 20 and 36 weeks pregnancy and 3 months post partum
  insulin resistance
Gestational diabetes | 18 months postpartum
  Insulin resistance

SECONDARY OUTCOMES:
incontinence | 20 and 36 weeks of pregnancy, 3 months post partum
  Fecal- and urinary incontinence (incontinence scores)
lumbopelvic pain | 20 and 36 weeks pregnancy and 3 months post partum
  Lumbopelvic pain (Pain intensity 100mm Visual Analogue Scale)
disability | 20 and 36 weeks pregnancy and 3 months post partum
  Disability Rating Index (Salèn et al. 1994)
incontinence | 18 months postpartum
  Fecal- and urinary incontinence (incontinence scores)
lumbopelvic pain | 18 months postpartum
  Lumbopelvic pain (Pain intensity 100mm Visual Analogue Scale)
disability | 18 months postpartum
  Disability Rating Index (Salèn et al. 1994)
Gestational diabetes | 5 years
  insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Siv Mørkved, PhD, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Department of Community Medicine and General Practice, Norwegian University of Science and Technology and Clinical Service, St Olavs Hospital, Trondheim University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Stafne SN, Salvesen KA, Romundstad PR, Eggebo TM, Carlsen SM, Morkved S. Regular exercise during pregnancy to prevent gestational diabetes: a randomized controlled trial. Obstet Gynecol. 2012 Jan;119(1):29-36. doi: 10.1097/AOG.0b013e3182393f86. PMID 22183208
- [Result] Stafne SN, Salvesen KA, Romundstad PR, Stuge B, Morkved S. Does regular exercise during pregnancy influence lumbopelvic pain? A randomized controlled trial. Acta Obstet Gynecol Scand. 2012 May;91(5):552-9. doi: 10.1111/j.1600-0412.2012.01382.x. Epub 2012 Mar 29. PMID 22364387
- [Result] Gustafsson MK, Stafne SN, Romundstad PR, Morkved S, Salvesen K, Helvik AS. The effects of an exercise programme during pregnancy on health-related quality of life in pregnant women: a Norwegian randomised controlled trial. BJOG. 2016 Jun;123(7):1152-60. doi: 10.1111/1471-0528.13570. Epub 2015 Aug 12. PMID 26265465
- [Result] Gustafsson MK, Romundstad PR, Stafne SN, Helvik AS, Stunes AK, Morkved S, Salvesen KA, Thorsby PM, Mosti MP, Syversen U. The effect of an exercise program in pregnancy on vitamin D status among healthy, pregnant Norwegian women: a randomized controlled trial. BMC Pregnancy Childbirth. 2019 Feb 20;19(1):76. doi: 10.1186/s12884-019-2220-z. PMID 30786861
- [Result] Johannessen HH, Froshaug BE, Lysaker PJG, Salvesen KA, Lukasse M, Morkved S, Stafne SN. Regular antenatal exercise including pelvic floor muscle training reduces urinary incontinence 3 months postpartum-Follow up of a randomized controlled trial. Acta Obstet Gynecol Scand. 2021 Feb;100(2):294-301. doi: 10.1111/aogs.14010. Epub 2020 Oct 30. PMID 32996139
- [Derived] Nyen SL, Stunes AK, Evensen KAI, Borsting T, Syversen U, Salvesen KA, Morkved S, Stafne SN. Associations between maternal and offspring glucose metabolism: a 9-year follow-up of a randomised controlled trial. Front Endocrinol (Lausanne). 2024 Jan 10;14:1324925. doi: 10.3389/fendo.2023.1324925. eCollection 2023. PMID 38269252
- [Derived] Bjontegaard KA, Stafne SN, Morkved S, Salvesen KA, Evensen KAI. Body mass index and physical activity in seven-year-old children whose mothers exercised during pregnancy: follow-up of a multicentre randomised controlled trial. BMC Pediatr. 2021 Nov 8;21(1):496. doi: 10.1186/s12887-021-02952-1. PMID 34743682
- [Derived] Stokkeland LMT, Giskeodegard GF, Ryssdal M, Jarmund AH, Steinkjer B, Madssen TS, Stafne SN, Stridsklev S, Lovvik TS, Iversen AC, Vanky E. Changes in Serum Cytokines Throughout Pregnancy in Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2022 Jan 1;107(1):39-52. doi: 10.1210/clinem/dgab684. PMID 34529073
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Derived] Stafne SN, Vollestad NK, Morkved S, Salvesen KA, Stendal Robinson H. Impact of job adjustment, pain location and exercise on sick leave due to lumbopelvic pain in pregnancy: a longitudinal study. Scand J Prim Health Care. 2019 Jun;37(2):218-226. doi: 10.1080/02813432.2019.1608058. Epub 2019 May 6. PMID 31057021
- [Derived] Hellenes OM, Vik T, Lohaugen GC, Salvesen KA, Stafne SN, Morkved S, Evensen KA. Regular moderate exercise during pregnancy does not have an adverse effect on the neurodevelopment of the child. Acta Paediatr. 2015 Mar;104(3):285-91. doi: 10.1111/apa.12890. Epub 2015 Feb 4. PMID 25471255
- [Derived] Helseth R, Salvesen O, Stafne SN, Morkved S, Salvesen KA, Carlsen SM. Gestational diabetes mellitus among Nordic Caucasian women: prevalence and risk factors according to WHO and simplified IADPSG criteria. Scand J Clin Lab Invest. 2014 Oct;74(7):620-8. doi: 10.3109/00365513.2014.928942. Epub 2014 Jul 1. PMID 24980704
- [Derived] Songoygard KM, Stafne SN, Evensen KAI, Salvesen KA, Vik T, Morkved S. Does exercise during pregnancy prevent postnatal depression? A randomized controlled trial. Acta Obstet Gynecol Scand. 2012 Jan;91(1):62-67. doi: 10.1111/j.1600-0412.2011.01262.x. Epub 2011 Oct 24. PMID 21880023